CLINICAL TRIAL: NCT04892277
Title: Phase I Dose Escalation Trial of CD19 Directed Chimeric Antigen Receptor T Cell Therapy in the Treatment of Relapsed/Refractory B Cell Malignancies
Brief Title: CD19-Directed CAR-T Cell Therapy for the Treatment of Relapsed/Refractory B Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC198A; NCI-2021-03969 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-007714 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-12; First posted 2021-05-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Specimen Handling; Biopsy; Cyclophosphamide; fludarabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cyclophosphamide, fludarabine, IC19/1563) (Experimental): Patients receive cyclophosphamide IV over 60 minutes and fludarabine IV over 30 minutes on days -5, -4, -3, or bendamustine IV over 10 minutes on days -4 and -3, and IC19/1563 IV on day 0. Patients also undergo bone marrow biopsy and aspiration, CT-PET or CT scans, MRI, and collection of blood and tissue samples throughout the trial.
  Interventions: Biological: Autologous Anti-CD19 CAR-expressing T-lymphocytes IC19/1563; Drug: Bendamustine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Autologous Anti-CD19 CAR-expressing T-lymphocytes IC19/1563 — Given IV
  Other Names: Autologous CAR-T Cells IC19/1563; CD19-directed CAR-T Cells IC19/1563; IC19 1563; IC19-1563; IC19/1563
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; Asta B 518; B-518; WR-138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo CT/PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial studies the effects of CD-19 directed chimeric antigen receptor (CAR)-T cell therapy for the treatment of patients with B cell malignancies that have come back (recurrent) or have not responded to treatment (refractory). CD-19 CAR-T cells use some of a patient's own immune cells, called T cells, to kill cancer. T cells fight infections and, in some cases, can also kill cancer cells. Some T cells are removed from the blood, and then laboratory, researchers will put a new gene into the T cells. This gene allows the T cells to recognize and possibly treat cancer. The new modified T cells are called the IC19/1563 treatment. IC19/1563 may help treat patients with relapsed/refractory B cell malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose of in-house, point of care manufactured autologous anti-CD19 CAR-expressing T-lymphocytes IC19/1563 (IC19/1563) in patient with relapsed/refractory B cell malignancies.

SECONDARY OBJECTIVES:

I. Assess the feasibility of in-house, point of care manufactured IC19/1563 cells.

II. Evaluate safety, including all grades of neurotoxicity (ICANS) and cytokine release syndrome as determined by the American Society for Transplantation and Cellular Therapy (ASTCT) criteria, by monitoring adverse events, laboratory abnormalities, vital signs, and other safety parameters.

III. Estimate the incidence of grade 3 or higher of neurotoxicity and cytokine release syndrome by grade 3 or higher neurotoxicity (ICANS) or CRS per the ASTCT criteria.

IV. Assess efficacy of a single dose of IC19/1563 cells:

IVa. Overall response rate (ORR); IVb. Duration of response (DOR); IVc. Progression-free survival (PFS); IVd. Minimal residual disease (MRD) negative bone marrow disease in patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), based on one month post evaluation.

CORRELATIVE RESEARCH OBJECTIVES:

I. Characterize the in vivo cellular kinetics profile (levels, persistence, trafficking) of CAR19 transgene and CD3+CAR+ cells into blood.

II. Characterize the changes in cytokine levels over time. III. Assess hospital resource utilization and health economics.

OUTLINE: This is a dose-escalation study of IC19/1563.

Patients receive cyclophosphamide intravenously (IV) over 60 minutes and fludarabine IV over 30 minutes on days -5, -4, -3, or bendamustine IV over 10 minutes on days -4 and -3, and IC19/1563 IV on day 0. Patients also undergo bone marrow biopsy and aspiration, computed tomography/positron emission tomography (CT/PET) or CT scans, magnetic resonance imaging (MRI), and collection of blood and tumor samples throughout the trial.

After completion of study treatment, patients are followed up on days 60, every 3 months up to year 3, every 6 months from years 3-5, and then annually for up to 15.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Relapsed or refractory CD19+ B cell malignancies of the one of the following histopathology:

  * Biopsy proven B-cell non-Hodgkin lymphoma (NHL) of any histopathology (including Richter Transformation of CLL); relapsed or refractory disease defined as:

    * Two or more prior lines of therapy, at least one anthracycline containing regimen, unless intolerable. Exception: Patients with Richter transformation of CLL are eligible if they had >= one prior treatment, including prior BTK inhibition
    * Demonstration of progressive or stable disease by positron emission tomography/computed tomography (PET/CT) or CT criteria as the best response to the most recent chemotherapy regimen according to the revised Lugano Response Criteria for Malignant Lymphoma.
    * Measurable disease defined as measurable by CT portion of a PET/CT: To be considered measurable, the must be at least one lesion that has a single diameter of (>1.5 cm Note: Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
  * Biopsy proven SLL or flow cytometry proven CLL; relapsed disease defined as:

    * >= two prior lines of therapy, and/or >= 6 months of second line prior BTK inhibition (e.g. venetoclax and ibrutinib). Exception: Patients in stable disease (SD) or partial response (PR) with a known ibrutinib resistance mutation (BTK or phospholipase Cgamma2) may be included even if on ibrutinib therapy for less than 6 months.
    * Demonstration of progressive or stable disease by PET/CT or CT criteria according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL2018) criteria
    * Measurable disease by CT portion of a PET/CT where at least one lesion has a single diameter of >1.5 cm or peripheral blood absolute blood lymphocyte count (ALC) of > 5000. Note: Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 8.0 g/dL (=< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 500/mm^3 (=< 14 days prior to registration)
* Platelet count >= 30,000/mm^3 (=< 14 days prior to registration)
* Total bilirubin =< 2.0 mg/dL (with the exception of subjects with Gilbert's syndrome. Subjects with Gilbert's syndrome may be included if their total bilirubin is =< 3.0 x upper limit of normal (ULN) and direct bilirubin =< 1.5 x ULN) (=< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 14 days prior to registration)
* Prothrombin time (PT) / international normalized ratio (INR) and/or activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (for patients receiving anticoagulation, there should be no prior history of bleeding, and no recent deep venous thrombosis/pulmonary embolism (DVT/PE) within the last 6 months of enrollment) (=< 14 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (=< 14 days prior to registration)
* Cardiac ejection fraction >= 50% and no evidence of clinically significant pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition scan (MUGA) scan
* Baseline oxygen saturation >= 92% on room air
* Negative serum pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Women patients of child bearing potential, including women with tubal ligations, must commit to using use 2 highly effective forms of birth control (defined as the use of an intrauterine device, a barrier method with spermicide, condoms, any form of hormonal contraceptives) for the duration of the study and for 12 months following IC19/1563 therapy
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Women of childbearing potential who are unwilling to employ highly effective contraception
* Sexually active males who are not willing to use contraception during the study and for >= 12 months after IC19/1563 therapy
* Patients who are able to obtain market approved CD19 CAR T-cell therapies
* Live vaccine =< 6 weeks prior to start of registration
* Autologous stem cell transplant =< 6 weeks of registration
* History of allogenic stem cell transplant if was performed less than 100 days prior to registration, if patients have active graft-versus host disease (GVHD) or are if patients are on chronic immunosuppression. Patients with allogeneic transplantation more than 100 days prior to registration, with no active GVHD and who are not on immunosuppression are eligible
* History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with central nervous system (CNS) involvement
* Any form of primary immunodeficiency such as severe combined immunodeficiency disease
* Current need of systemic corticosteroid therapy, in doses over 20 mg /day of prednisone or equivalent forms of steroids
* History of severe immediate hypersensitivity reaction to CART19, stem cell infusion dimethyl sulfoxide (DMSO) or any of the CAR-T cryopreservation ingredients
* History of malignancy other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast) or early stage cancers (Stage I or II), unless disease free for >= 2 years
* Clinically significant active infection (e.g. simple urinary tract infection [UTI], bacterial pharyngitis allowed) or currently receiving IV antibiotics or have received IV antibiotics =< 7 days prior to registration. Note: prophylactic antibiotics, antivirals and antifungals are permitted
* Known history of human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or hepatitis C infection. Subjects with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines. Prophylactic antiviral therapy should be considered per institutional guidelines
* History of any of the following cardiovascular conditions =< 6 months:

  * Class III or IV heart failure as defined by the New York Heart Association (NYHA)
  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Or other clinically significant cardiac disease
* Any other acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or that, in the judgment of the investigator, would make the subject inappropriate for entry into the study
* Concurrent cancer therapy. The following are exceptions:

  * Treatment with therapies may continue at time of registration; however, the washout period must be met prior to leukapheresis
  * Treatment with any other investigational agent may continue at time of registration provided last date of treatment is =< 14 days prior to leukapheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2028-03-27 (Estimated); Study Completion 2040-03-27 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 90 days
  MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients).

SECONDARY OUTCOMES:
Proportion of patients who achieve a successful infusion without manufacturing failure or out of spec products | Up to 15.5 years
  All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for assessing feasibility. Exact binomial 95% confidence intervals for the true rate of successful infusion will be calculated.
Overall response rate (ORR) | From a complete response (CR) or partial response (PR) noted as the objective status at any time after the start of CART19 infusion, assessed up to 15.5 years
  ORR will be estimated by the number of patients who achieve a response divided by the total number of evaluable patients who have received a successful chimeric antigen receptor (CAR)-T19 infusion. Response criteria will follow the revised International working group Response Criteria for Malignant Lymphoma or the 2018 International Workshop for Chronic Lymphocytic Leukemia (CLL) response criteria. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Duration of response (DOR) | From CR or PR to the date of progression or death, assessed up to 15.5 years
  The distribution of duration of response will be estimated using the method of Kaplan Meier.
Progression-free survival | From registration to disease progression or death, assessed up to 15.5 years
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Rates of grade 3 or higher neurotoxicity | Up to 15.5 years
  Assessed per American Society for Transplantation and Cellular Therapy (ASTCT) guidelines will be estimated by the number of patients who experience grade 3 or higher of neurotoxicity divided by the total number of evaluable patients. Assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. In addition, neurotoxicity will be assessed by Immune Effector Cell Associated Neurotoxicity Syndrome criteria. Exact binomial 95% confidence intervals for the true rates of grade 3 or higher neurotoxicity will be calculated.
Rate of cytokine release syndrome | Up to 15.5 years
  Assessed per ASTCT guidelines will be estimated by the number of patients who experience cytokine release syndrome divided by the total number of evaluable patients. Cytokine release syndrome will be evaluated by CTCAE version 5.0 and Lee grading criteria. Exact binomial 95% confidence intervals will be used.
Minimal residual disease (MRD) | 1 month
  MRD negative rate will be estimated by the number of CLL/small lymphocytic lymphoma (SLL) patients with MRD negative bone marrow divided by the total number of evaluable CLL/SLL patients. Exact binomial 95% confidence intervals for the true rate of MRD negativity will be calculated.

OTHER OUTCOMES:
In vivo cellular kinetics profile of CAR19 cells | Up to 15.5 years
  The in vivo cellular kinetics profile (levels, persistence, trafficking) of CAR19 transgene and CD3+CAR+ cells into blood will be summarized descriptively. This will include levels of CAR19 transgene by real time polymerase chain reaction in blood and bone marrow and levels of CART19 detected by flow cytometry in blood.
Serum/plasma levels of cytokines | Baseline up to 30 days
  Will be monitored at baseline and at multiple time points after CART19 infusion. Values at each time point and changes across time will be summarized graphically and descriptively.
The total number of hospitalizations and ICU admissions | Up to 15.5 years
  These measures will be summarized descriptively.
Length of stay in hospital | Up to 15.5 years
  These measures will be summarized descriptively.
Time between cell collection and infusion | Up to 15.5 years
  These measures will be summarized descriptively.
Total cost of product | Up to 15.5 years
  These measures will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Saad J. Kenderian, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials